CLINICAL TRIAL: NCT06807840
Title: Evaluating Immune Imprinting in the Context of Influenza Virus Infections
Brief Title: Flu Infection at UPHS
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 857436; 75N93021C00015-P00012-9999-1 (NIH)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Influenza Human
Keywords: Flu Infection at UPHS
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: influenza virus infection — Participants with active influenza virus infection will be enrolled in this study.

SUMMARY:
Cellular and humoral immune responses in individuals with active influenza infection will be assessed. Each year, up to 50 participants will be enrolled. The investigators hypothesize that influenza infection will elicit mostly memory immune responses rather than de novo immune responses to infection.

DETAILED DESCRIPTION:
Using samples collected from individuals after influenza virus vaccination, the investigators have shown that immune cells primed by previous influenza exposures are recruited to produce antibodies against newer viral strains. The investigators previous work indicate that the majority of the immune cells that respond to influenza vaccination are from the memory compartment, suggesting that 'immune imprinting' greatly affects the specificity of antibodies elicited by influenza vaccines. It remains less clear how prior influenza virus exposures impact immunity elicited by influenza virus infections. Compared to vaccinated individuals, it is more difficult to enroll influenza virus infected patients and track their immune responses over time. Viral antigens can persist for longer amounts of time following influenza virus infections relative to influenza vaccinations. It is therefore possible that influenza virus infections more efficiently prime de novo immune responses compared to influenza virus vaccinations. In this study, the investigators will longitudinally collect serum, PBMC, and respiratory samples from influenza virus-infected individuals from the University of Pennsylvania Health System characterize the cellular and humoral immune responses elicited by influenza virus infections.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Aged 18 years and older
4. Influenza positive test result performed within the University of Pennsylvania Health System

Exclusion Criteria:

1. Known latex allergy
2. Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months
3. Pregnancy due to the volume of blood collected in this study
4. Treatment with immunoglobulin or another blood product within the 3 months prior to enrollment in this study
5. Any neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy ("active" is defined as having received treatment within the past 5 years)
6. Known acute or chronic medical condition that, in the opinion of the investigator or appropriate sub-investigator, would interfere with the evaluation of immune responses
7. Intends to donate blood during the study period
8. A known human immunodeficiency virus, hepatitis B, or hepatitis C infection
9. Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
10. Prolonged inpatient hospitalization that disrupts or interferes with study procedures.
11. Weigh less than 110lbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 50 influenza virus-infected participants who have tested positive for influenza virus infection within the University of Pennsylvania Health System will be enrolled in the study. Potential candidates will be in the Emergency Department with influenza-like symptoms and will be eligible once the eligibility criteria are met.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Effect of influenza virus infection on neutralizing antibody titers to contemporary and historical influenza virus strains | 2 years
  The investigators will compare neutralizing antibodies in sera, plasma, and nasal swab samples against the influenza strain that each participant is infected with as well as historical and recently circulating influenza virus strains. Antibody titers between different strains will be compared to understand if memory or de novo immune responses are generated following influenza infection based on inferred influenza exposure history.

SECONDARY OUTCOMES:
Differences in binding antibodies against historical and contemporary influenza virus strains in individuals following influenza virus infection | 2 years
  The investigators will compare binding antibodies in sera, plasma, and nasal swab samples against the influenza strain that each participant is infected with as well as historical and recently circulating influenza virus strains. Antibody titers between different strains will be compared to understand if memory or de novo immune responses are generated following influenza infection based on inferred influenza exposure history.
Characterize B cell responses to influenza following influenza virus infection | 2 years
  Influenza specific B cells will be identified in PBMC samples and their specificity and functionality to different influenza virus strains will be assessed to understand how influenza infection influences the generation of memory and de novo immune responses.
Characterize T cell responses to influenza following influenza virus infection | 2 years
  T cells specific to influenza will be identified in PBMC samples and their specificity and functionality to different influenza virus strains will be assessed to understand how influenza infection influences the generation of memory and de novo immune responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol and statistical analysis plan may need to be shared for publication.
Supporting Information: Study Protocol, SAP
Time Frame: At publication
Access Criteria: Per journal publication policy